CLINICAL TRIAL: NCT07354711
Title: A Phase I/II Study of 3H-10000 (an Anti-FGFR2b Antibody-Drug Conjugate) in Subjects With Unresectable or Metastatic Advanced Solid Tumors
Brief Title: A First-in-human Study of 3H-10000 in Patients With Unresectable or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: 3H Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3H-10000-101
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer; Stomach Cancer
MeSH Terms: conditions — Lung Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stage I - dose escalation (Experimental): Dose escalation of 3H-10000 in patients with advanced solid tumors.
  Interventions: Drug: 3H-10000
- stage II - expansion (Experimental): Expansion evaluating the recommended dose and schedule of 3H-10000 identified from Stage I.
  Interventions: Drug: 3H-10000

INTERVENTIONS:
Drug: 3H-10000 — 3H-10000 will be administered by infusion Q2W in 28-day cycles.

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, efficacy, pharmacokinetics, and pharmacodynamics of 3H-10000 in the treatment of unresectable or metastatic solid tumors .

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing and able to sign the ICF and to adhere to the study visit schedule and other protocol requirements.
* Male or female subjects aged ≥18 years at the time of signing the ICF.
* According to RECIST v1.1, there is at least one measurable lesion.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1 point.
* Life expectancy of ≥3 months.

Exclusion Criteria:

* Meningeal diseases or carcinomatous meningitis.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage every two weeks or more frequently.
* Having received treatment with other investigational drugs within 4 weeks prior to the first dose of the study drug.
* Any AEs induced by prior anti-tumor therapy having not resolved to Grade 1 or lower (except for alopecia or any other Grade 2 AEs assessed by the investigator as not being associated with any safety risk).
* Any corneal or retinal disease/keratopathy assessed by the investigator as of clinical significance, including but not limited to bullous/band keratopathy, corneal abrasion, inflammation/ulceration, and keratoconjunctivitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2026-01-04 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Phase：Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 2 years
  Number of participants with AEs and SAEs as graded by the National Cancer Institute- Common Terminology Criteria for Adverse Events Version (NCI CTCAE 5.0)), including AEs that meet protocol-defined dose-limiting toxicity (DLT) criteria and AEs meeting protocol-defined adverse event of clinical interest (AECIs)
Dose Escalation Phase：Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of 3H-10000 | Up to approximately 2 years
  The MTD or MAD is defined as the highest dose evaluated for which the estimated toxicity rate is closest to a target toxicity rate, or the highest dose administered, respectively.
Dose Escalation Phase：The recommended Phase 2 dose (RP2D) of 3H-10000 | Up to approximately 2 years
  The RP2D of 3H-10000 monotherapy will be determined based on relevant data, as available
Efficacy Expansion Phase：Overall Response Rate (ORR) | Up to approximately 2 years
  ORR is defined as the percentage of participants with confirmed complete response (CR) or partial response (PR) by Response Evaluations Criteria in Solid Tumors Version 1.1 (RECIST v1.1)

SECONDARY OUTCOMES:
Dose Escalation Phase：ORR | Up to approximately 2 years
  ORR is defined as the percentage of participants with CR or PR, as determined by RECIST v1.1
Dose Escalation Phase and Efficacy Expansion Phase：Disease Control Rate (DCR) | Up to approximately 2 years
  DCR is defined as the percentage of participants with best overall response of a CR, PR, and stable disease, as assessed by RECIST v1.1
Dose Escalation Phase and Efficacy Expansion Phase：Duration of Response (DOR) | Up to approximately 2 years
  DOR is defined as the time from the first determination of an objective response per RECIST v1.1 until the first documentation of progression or death, whichever comes first, as assessed using RECIST v1.1
Efficacy Expansion Phase：Progression Free Survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the date of the first dose of study drug to the date of the first documentation of progressive disease assessed using RECIST v1.1 or death, whichever occurs first
Efficacy Expansion Phase：Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 2 years
  Number of participants with AEs and SAEs as graded by the National Cancer Institute- Common Terminology Criteria for Adverse Events Version (NCI CTCAE 5.0), and AEs meeting protocol-defined adverse event of clinical interest (AECI)s.
Dose Escalation Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Twice in the first 3 months
  AUC0-last
Dose Escalation Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Twice in the first 3 months
  AUC0-inf
Dose Escalation Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Twice in the first 3 months
  Cmax
Dose Escalation Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Twice in the first 3 months
  Tmax
Dose Escalation Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Twice in the first 3 months
  Ctrough
Dose Escalation Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Twice in the first 3 months
  CL
Dose Escalation Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Twice in the first 3 months
  t1/2
Dose Escalation Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Twice in the first 3 months
  Vd
Dose Escalation Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Twice in the first 3 months
  Vss
Efficacy Expansion Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Up to approximately 2 years
  AUC0-last
Efficacy Expansion Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Up to approximately 2 years
  AUC0-inf
Efficacy Expansion Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Up to approximately 2 years
  Cmax
Efficacy Expansion Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Up to approximately 2 years
  Tmax
Efficacy Expansion Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Up to approximately 2 years
  Ctrough
Efficacy Expansion Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Up to approximately 2 years
  CL
Efficacy Expansion Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Up to approximately 2 years
  t1/2
Efficacy Expansion Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Up to approximately 2 years
  Vd
Efficacy Expansion Phase：To evaluate the pharmacokinetics (PK) of 3H-10000 | Up to approximately 2 years
  Vss

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China